CLINICAL TRIAL: NCT02173704
Title: A Phase 3, Open Label, Randomized, Controlled, Multi-Center Study to Evaluate the Safety and Immunogenicity of GSK Biologicals' Meningococcal B Recombinant Vaccine When Administered Concomitantly With Routine Vaccines to Healthy Infants in Taiwan.
Brief Title: Safety and Immunogenicity of GlaxoSmithKline (GSK) Biologicals' Meningococcal B Recombinant Vaccine When Administered Concomitantly With Routine Vaccines to Healthy Infants of 2 Months of Age and Older, in Taiwan.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 205249; V72_60 (Other: Novartis); 2014-005568-14 (EudraCT Number)
Record Dates: First submitted 2014-06-05; First posted 2014-06-25 (Estimated); Results first posted 2018-06-15 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Meningococcal Disease; Infections, Meningococcal
Keywords: Meningitis; Infants; Meningococcal B Recombinant Vaccine
MeSH Terms: conditions — Meningococcal Infections; Meningitis | interventions — 4CMenB vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bexsero + Routine Group (Experimental): Subjects received three doses of Bexsero® vaccine at 2, 4, 6 months followed by a booster dose at 12 months, concomitantly administered with routine vaccines (i.e. combined Infanrix-IPV + Hib® and Prevenar-13® at 2, 4, 6 months of age; Engerix-B® at 6 months of age; Priorix® and Varilrix® at 12 months of age.
  Interventions: Biological: Bexsero®
- Routine Group (Active Comparator): Subjects received routine vaccines Infanrix-IPV + Hib® and Prevenar-13® at 2, 4, 6 months of age; Engerix-B® vaccine at 6 months; Priorix® and Varilrix® vaccines at 12 months of age.
  Interventions: Biological: Routine vaccines

INTERVENTIONS:
Biological: Bexsero® — Four doses administered in the anterolateral area of the right or left thigh.
  Arms: Bexsero + Routine Group
Biological: Routine vaccines — Infanrix-IPV + Hib®, Prevenar-13®, Engerix-B®, Priorix® and Varilrix® administered in the anterolateral area of the right or left thigh.
  Arms: Routine Group

SUMMARY:
Assess the safety and immunogenicity of a 3-dose schedule (at 2, 4, 6 months) of GSK Biologicals' Meningococcal B recombinant vaccine followed by a booster at 12 months when concomitantly administered with routine vaccines in healthy infants in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

1. healthy 2-month old infants (55-89 days, inclusive), who were born after full term pregnancy with an estimated gestational age ≥ 37 weeks and a birth weight ≥ 2.5 kg;
2. for whom a parent/legal guardian has given written informed consent after the nature of the study has been explained;
3. available for all the visits scheduled in the study;
4. in good health as determined by medical history, physical examination and clinical judgment of the investigator.

Exclusion Criteria:

1. History of any meningococcal vaccine administration;
2. Prior vaccination with any Diphtheria, Tetanus, Pertussis (acellular or whole cell), Polio (either Inactivated or Oral), Haemophilus influenzae type b (Hib), Pneumococcal, MMR or varicella antigens;
3. Previous ascertained or suspected disease caused by N. meningitidis;
4. Household contact with and/or intimate exposure to an individual with laboratory confirmed N. meningitidis;
5. History of severe allergic reaction after previous vaccinations or hypersensitivity to any vaccine component;
6. Significant acute or chronic infection within the previous 7 days or body temperature higher or equal to 38C degrees within the previous day;
7. Antibiotics within 6 days prior to enrollment;
8. Any serious chronic or progressive disease according to the judgment of the investigator (e.g., neoplasm, insulin dependent diabetes mellitus Type I, cardiac disease, hepatic disease, progressive neurological disease or seizure, either associated with fever or as part of an underlying neurological disorder or syndrome, autoimmune disease, HIV infection or AIDS, or blood dyscrasias or diathesis, signs of cardiac or renal failure or severe malnutrition);
9. Known or suspected impairment/alteration of the immune system, immunosuppressive therapy, use of systemic corticosteroids or chronic use of inhaled high-potency corticosteroids since birth;
10. Receipt of blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation;
11. Receipt of, or intent to immunize with any other vaccine(s) (with the exception of rotavirus vaccine, influenza vaccine and second HepB vaccine), within 28 days prior and throughout the study period. Furthermore, subjects must have received HepB vaccine preferably at 0, 1 month of age, with the second dose at least 14 days prior to study vaccination. Influenza vaccine should be administered at least 14 days before or 14 days after study vaccination; Rotavirus vaccine may be administered during the study as per local practice.
12. Participation in another clinical trial since birth or planned for during study;
13. Family members and household members of research staff;
14. Any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.

Ages: 55 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 225 (Actual)
Dates: Start 2014-09-11 (Actual); Primary Completion 2015-12-25 (Actual); Study Completion 2016-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Background] Chiu NC, Huang LM, Willemsen A, Bhusal C, Arora AK, Reynoso Mojares Z, Toneatto D. Safety and immunogenicity of a meningococcal B recombinant vaccine when administered with routine vaccines to healthy infants in Taiwan: A phase 3, open-label, randomized study. Hum Vaccin Immunother. 2018 May 4;14(5):1075-1083. doi: 10.1080/21645515.2018.1425659. Epub 2018 Feb 15. PMID 29337653
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 2 sites in Taiwan
Pre-assignment Details: All subjects were enrolled
Period: Overall Study
Arm/Group | Bexsero + Routine Group | Routine Group
Started | 150 | 75
Completed | 137 | 71
Not Completed | 13 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bexsero + Routine Group | Routine Group | Total
Number analyzed (Participants) | 150 | 75 | 225
Age, Continuous [Mean (Standard Deviation); unit: Days] | 67.9 (6.46) | 68.9 (6.86) | 68.3 (6.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 27 | 109
  Male | 68 | 48 | 116

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Human Serum Bactericidal Activity (hSBA) Titer ≥ 1:5 Against Neisseria Meningitidis Serogroup B Strains
Description: Percentage of subjects with hSBA titer ≥ 1:5 at 1 month following the third vaccination (at 7 months of age) against the indicator strains H44/76, 5/99, NZ98/254 and strain M10713 when Bexsero® was given concomitantly with routine vaccines (Infanrix-IPV + Hib®, Prevenar-13® and Engerix-B®).
Time Frame: At Day 1 and at one month after the third vaccination (Day 152)
Population: Analysis was done on Full Analysis Population (FAS) population day 152, which included all subjects in the exposed set who received at least one dose of a study vaccination and provided immunogenicity data at relevant time points.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | Bexsero + Routine Group | Routine Group
Number analyzed (Participants) | 135 | 71
Percentages of subjects
  H44/76 strain [Day 1]: number analyzed (Participants) | 116 | 59
  H44/76 strain [Day 1] | 0 [0.0 to 3.1] | 0 [0.0 to 6.1]
  H44/76 strain [Day 152]: number analyzed (Participants) | 130 | 66
  H44/76 strain [Day 152] | 100 [97.2 to 100] | 0 [0.0 to 5.4]
  5/99 strain [Day 1]: number analyzed (Participants) | 124 | 69
  5/99 strain [Day 1] | 1 [0.02 to 4.4] | 1 [0.04 to 7.8]
  5/99 strain [Day 152]: number analyzed (Participants) | 129 | 70
  5/99 strain [Day 152] | 100 [97.2 to 100] | 0 [0.0 to 5.1]
  M10713 strain [Day 1]: number analyzed (Participants) | 100 | 57
  M10713 strain [Day 1] | 10 [4.9 to 17.6] | 19 [10 to 31.9]
  M10713 strain [Day 152]: number analyzed (Participants) | 123 | 65
  M10713 strain [Day 152] | 59 [50.1 to 68.1] | 8 [2.5 to 17]
  NZ98/254 strain [Day 1]: number analyzed (Participants) | 134 | 71
  NZ98/254 strain [Day 1] | 0 [0.0 to 2.7] | 0 [0.0 to 5.1]
  NZ98/254 strain [Day 152] | 79 [71.4 to 85.8] | 0 [0.0 to 5.1]
Statistical Analysis 1: Comparison: Bexsero + Routine Group vs Routine Group; Statistical analysis 5/99 strain: The power to reject the null hypothesis associated with the primary objective for strain 5/99 was 99%; Test type: Non-Inferiority or Equivalence — Sufficiency: The criterion for a sufficient immune response was that the lower limit of the two-sided 95% CI for the percentage of subjects with hSBA titer ≥1:5 should be ≥ 70%; Exact test of binomial proportion; Single binomial proportion = 100, 95% CI 2-sided [97.2 to 100]
Statistical Analysis 2: Comparison: Bexsero + Routine Group vs Routine Group; Statistical analysis NZ98/254 strain: The power to reject the null hypothesis associated with the primary objective for strain NZ98/25 was 94%; Test type: Non-Inferiority or Equivalence — Sufficiency: The criterion for a sufficient immune response was that the lower limit of the two-sided 95% CI for the percentage of subjects with hSBA titer ≥ 1:5 should be ≥ 70%; Exact test of binomial proportion; single binomial proportion = 79, 95% CI 2-sided [71.4 to 85.8]

2. Primary Outcome: Percentage of Subjects With Human Serum Bactericidal Assay (hSBA) Titer ≥ 1:4 Against Neisseria Meningitidis Serogroup B Strains
Description: Percentage of subjects with hSBA titer ≥ 1:4 at 1 month after third vaccination (at 7 months of age) against the indicator strains H44/76, 5/99, NZ98/254 and strain M10713 when Bexsero® was given concomitantly with routine vaccines (Infanrix-IPV + Hib®, Prevenar-13® and Engerix-B®).
Time Frame: At Day 1 and at one month after third vaccination (Day 152)
Population: Analysis was done on Full Analysis Set (FAS) population day 152. The FAS population included all subjects in the exposed set who received at least one dose of a study vaccination and provided immunogenicity data at relevant time points.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Bexsero + Routine Group | Routine Group
Number analyzed (Participants) | 136 | 71
Percentage of subjects
  H44/76 strain [Day 1]: number analyzed (Participants) | 116 | 59
  H44/76 strain [Day 1] | 0 [0.0 to 3.1] | 0 [0.0 to 6.1]
  H44/76 strain [Day 152]: number analyzed (Participants) | 130 | 66
  H44/76 strain [Day 152] | 100 [97.2 to 100] | 0 [0.0 to 5.4]
  5/99 strain [Day 1]: number analyzed (Participants) | 124 | 69
  5/99 strain [Day 1] | 1 [0.02 to 4.4] | 1 [0.04 to 7.8]
  5/99 strain [Day 152]: number analyzed (Participants) | 129 | 70
  5/99 strain [Day 152] | 100 [97.2 to 100] | 0 [0.0 to 5.1]
  M10713 strain [Day 1]: number analyzed (Participants) | 100 | 57
  M10713 strain [Day 1] | 11 [5.6 to 18.8] | 25 [14.1 to 37.8]
  M10713 strain [Day 152]: number analyzed (Participants) | 123 | 65
  M10713 strain [Day 152] | 71 [61.9 to 78.6] | 8 [2.5 to 17.0]
  NZ98/254 strain [Day 1]: number analyzed (Participants) | 134 | 71
  NZ98/254 strain [Day 1] | 0 [0.0 to 2.7] | 0 [0.0 to 5.1]
  NZ98/254 strain [Day 152]: number analyzed (Participants) | 135 | 71
  NZ98/254 strain [Day 152] | 87 [80.6 to 92.5] | 0 [0.0 to 5.1]

3. Secondary Outcome: Percentage of Subjects With hSBA Titer ≥ 1:5 Against Neisseria Meningitidis Serogroup B, When Bexsero® Booster Was Given With Routine Vaccines (Priorix® + Varilrix® Vaccines)
Description: Percentage of subjects with hSBA titer ≥ 1:5 before booster vaccination and after booster vaccination when Bexsero® booster dose was given with routine vaccines (Priorix® + Varilrix® vaccine) as compared to when only routine vaccines were administered.
Time Frame: At Day 305 and Day 335
Population: Analysis was done on FAS population Day 335. The FAS population included all subjects in the exposed set who received at least one dose of a study vaccination and provided immunogenicity data at relevant time points.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Bexsero + Routine Group | Routine Group
Number analyzed (Participants) | 136 | 71
Percentage of subjects
  H44/76 strain [Day 305]: number analyzed (Participants) | 123 | 64
  H44/76 strain [Day 305] | 81 [73.3 to 87.8] | 2 [0.04 to 8.4]
  H44/76 strain [Day 335]: number analyzed (Participants) | 127 | 64
  H44/76 strain [Day 335] | 99 [95.7 to 99.98] | 2 [0.04 to 8.4]
  5/99 strain [Day 305]: number analyzed (Participants) | 135 | 70
  5/99 strain [Day 305] | 99 [94.8 to 99.82] | 1 [0.04 to 7.7]
  5/99 strain [Day 335]: number analyzed (Participants) | 134 | 71
  5/99 strain [Day 335] | 99 [94.7 to 99.82] | 0 [0 to 5.1]
  M10713 strain [Day 305]: number analyzed (Participants) | 130 | 65
  M10713 strain [Day 305] | 22 [14.8 to 29.6] | 11 [4.4 to 20.9]
  M10713 strain [Day 335]: number analyzed (Participants) | 130 | 69
  M10713 strain [Day 335] | 92 [86.3 to 96.2] | 13 [6.1 to 23.3]
  NZ98/254 strain [Day 305]: number analyzed (Participants) | 136 | 70
  NZ98/254 strain [Day 305] | 17 [11 to 24.3] | 1 [0.04 to 7.7]
  NZ98/254 strain [Day 335] | 94 [88.7 to 97.4] | 0 [0 to 5.1]
Statistical Analysis 1: Comparison: Bexsero + Routine Group vs Routine Group; Statistical analysis H44/76 strain: The null hypothesis associated with the primary objective is that the proportion of subjects with hSBA titers ≥ 1:5 one month after the third dose of the Bexsero® vaccine was ≤ 0.70. Assuming the results for the three strains are independent, the power to reject the null hypothesis associated with the primary objectives to demonstrate sufficiency of response (for all three strains was 92%; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Exact test of binomial proportion; Single binomial proportion = 99, 95% CI 2-sided [95.7 to 99.98]
Statistical Analysis 2: Comparison: Bexsero + Routine Group vs Routine Group; Statistical analysis 5/99 strain: The power to reject the null hypothesis associated with the secondary objective for strain 5/99 was 99%; Test type: Non-Inferiority or Equivalence — Sufficiency: The criterion for a sufficient immune response was that the lower limit of the two-sided 95% CI for the percentage of subjects with hSBA titer ≥1:5 should be ≥ 75%; Exact test for binomial proportion; Single binomial proportion = 99, 95% CI 2-sided [94.7 to 99.82]
Statistical Analysis 3: Comparison: Bexsero + Routine Group vs Routine Group; Statistical analysis NZ98/254 strain: The power to reject the null hypothesis associated with the secondary objective for strain NZ98/254 was 99%; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 2]; Exact test for binomial proportions; Single binomial proportion = 94, 95% CI 2-sided [88.7 to 97.4]

4. Secondary Outcome: hSBA Geometric Mean Titers (GMTs) Against Neisseria Meningitidis Serogroup B Indicator Strains, When Bexsero® Vaccine Was Given With Routine Vaccines
Description: hSBA GMTs against the indicator strains H44/76, 5/99, NZ98/254 and strain M10713 was evaluated at baseline (2 months of age, Day 1), 1 month after the third vaccination with Bexsero® with concomitant routine vaccines (Infanrix-IPV+Hib®, Prevenar-13®, Engerix®) (7 months of age, Day 152) or prior to the booster dose of Bexsero® with routine vaccines (Priorix®, Varilrix®) (12 months of age, Day 305) and 1 month after the booster dose (13 months of age, Day 335), as compared to when only routine vaccines were administered.
Time Frame: At Day 1, Day 152, Day 305 and Day 335
Population: Analysis was performed on the FAS population, which included all subjects in the exposed set who received at least one dose of a study vaccination and provided immunogenicity data at relevant time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Bexsero + Routine Group | Routine Group
Number analyzed (Participants) | 145 | 73
Titer
  H44/76 strain [Day 1]: number analyzed (Participants) | 132 | 65
  H44/76 strain [Day 1] | 1.01 [0.99 to 1.02] | 1.02 [0.98 to 1.05]
  H44/76 strain [Day 152]: number analyzed (Participants) | 130 | 66
  H44/76 strain [Day 152] | 72 [64 to 81] | 1.01 [0.99 to 1.03]
  H44/76 strain [Day 305]: number analyzed (Participants) | 123 | 64
  H44/76 strain [Day 305] | 11 [9.27 to 13] | 1.26 [1.06 to 1.5]
  H44/76 strain [Day 335]: number analyzed (Participants) | 127 | 64
  H44/76 strain [Day 335] | 157 [131 to 188] | 1.1 [1.01 to 1.19]
  5/99 strain [Day 1]: number analyzed (Participants) | 141 | 72
  5/99 strain [Day 1] | 1.08 [0.98 to 1.18] | 1.03 [0.98 to 1.08]
  5/99 strain [Day 152]: number analyzed (Participants) | 129 | 70
  5/99 strain [Day 152] | 963 [864 to 1073] | 1 [1 to 1]
  5/99 strain [Day 305]: number analyzed (Participants) | 135 | 70
  5/99 strain [Day 305] | 205 [174 to 242] | 1.1 [0.91 to 1.33]
  5/99 strain [Day 335]: number analyzed (Participants) | 134 | 71
  5/99 strain [Day 335] | 2315 [1893 to 2832] | 1 [1 to 1]
  M10713 strain [Day 1]: number analyzed (Participants) | 121 | 64
  M10713 strain [Day 1] | 1.36 [1.2 to 1.54] | 1.75 [1.37 to 2.24]
  M10713 strain [Day 152]: number analyzed (Participants) | 123 | 65
  M10713 strain [Day 152] | 8.41 [6.63 to 11] | 1.25 [1.08 to 1.46]
  M10713 strain [Day 305]: number analyzed (Participants) | 130 | 65
  M10713 strain [Day 305] | 2.18 [1.81 to 2.63] | 1.6 [1.34 to 1.91]
  M10713 strain [Day 335]: number analyzed (Participants) | 130 | 69
  M10713 strain [Day 335] | 17 [14 to 20] | 1.58 [1.33 to 1.89]
  NZ98/254 strain [Day 1] | 1.01 [0.99 to 1.02] | 1 [1 to 1]
  NZ98/254 strain [Day 152]: number analyzed (Participants) | 135 | 71
  NZ98/254 strain [Day 152] | 9.2 [7.82 to 11] | 1.02 [0.98 to 1.05]
  NZ98/254 strain [Day 305]: number analyzed (Participants) | 136 | 70
  NZ98/254 strain [Day 305] | 1.91 [1.63 to 2.25] | 1.04 [0.98 to 1.1]
  NZ98/254 strain [Day 335]: number analyzed (Participants) | 136 | 71
  NZ98/254 strain [Day 335] | 26 [21 to 31] | 1 [1 to 1]

5. Secondary Outcome: hSBA Geometric Mean Ratios (GMRs) Against Neisseria Meningitidis Serogroup B Strains.
Description: GMRs of post-vaccination versus pre-vaccination of hSBA titer against the indicator strains H44/76, 5/99, NZ98/254 and strain M10713 were evaluated at one month after the third vaccination with Bexsero® vaccine and concomitant routine vaccines (Infanrix-IPV+Hib®, Prevenar-13® and Engerix®) (Day 152) compared to baseline (Day 1) or at one month after the booster dose of Bexsero® vaccine with routine vaccines (Priorix®, Varilrix®) (Day 335) compared to prior to the booster dose (Day 305).
Time Frame: At Day 1, Day 152, Day 305 and Day 335
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Bexsero + Routine Group | Routine Group
Number analyzed (Participants) | 135 | 71
Ratio
  H44/76 strain [Day 152/Day 1]: number analyzed (Participants) | 116 | 59
  H44/76 strain [Day 152/Day 1] | 71 [63 to 80] | 0.99 [0.95 to 1.04]
  H44/76 strain [Day 335/Day 305]: number analyzed (Participants) | 113 | 56
  H44/76 strain [Day 335/Day 305] | 155 [127 to 188] | 1.07 [0.97 to 1.19]
  5/99 strain [Day 152/Day 1]: number analyzed (Participants) | 124 | 69
  5/99 strain [Day 152/Day 1] | 875 [752 to 1019] | 0.97 [0.93 to 1.03]
  5/99 strain [Day 335/Day 305]: number analyzed (Participants) | 129 | 70
  5/99 strain [Day 335/Day 305] | 2110 [1674 to 2659] | 0.97 [0.93 to 1.03]
  M10713 strain [Day 152/Day 1]: number analyzed (Participants) | 100 | 57
  M10713 strain [Day 152/Day 1] | 5.69 [4.25 to 7.61] | 0.68 [0.54 to 0.85]
  M10713 strain [Day 335/Day 305]: number analyzed (Participants) | 105 | 60
  M10713 strain [Day 335/Day 305] | 12 [8.99 to 15] | 0.91 [0.68 to 1.21]
  NZ98/254 strain [Day 152/Day 1]: number analyzed (Participants) | 134 | 71
  NZ98/254 strain [Day 152/Day 1] | 9.18 [7.79 to 11] | 1.02 [0.98 to 1.05]
  NZ98/254 strain [Day 335/Day 305] | 25 [21 to 31] | 1 [1 to 1]

6. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥1:8 Against Neisseria Meningitidis Serogroup B, When Bexsero® Vaccine Was Given With Routine Vaccines
Description: Percentages of subjects with hSBA titers ≥1:8 against N.meningitidis serogroup B strains, at one month after concomitant administration of third primary dose of Bexsero® with routine vaccines [Infanrix-IPV + Hib®, Prevenar-13® and Engerix-B®] and at one month after concomitant administration of Bexsero® booster dose with routine vaccines [Priorix® and Varilrix® vaccine],as compared to when only routine vaccines were administered.
Time Frame: At Day 1,Day 152,Day 305, Day 335
Population: Analysis was done on FAS population, which included all subjects in the exposed set who received at least one dose of a study vaccination and provided immunogenicity data at relevant time points.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | Bexsero + Routine Group | Routine Group
Number analyzed (Participants) | 145 | 73
Percentages of subjects
  H44/76 strain (Day 1): number analyzed (Participants) | 132 | 65
  H44/76 strain (Day 1) | 0 [0.0 to 2.8] | 0 [0.0 to 5.5]
  H44/76 strain (Day 152): number analyzed (Participants) | 130 | 66
  H44/76 strain (Day 152) | 100 [97.2 to 100] | 0 [0.0 to 5.4]
  H44/76 strain (Day 305): number analyzed (Participants) | 123 | 64
  H44/76 strain (Day 305) | 66 [56.8 to 74.2] | 2 [0.04 to 8.4]
  H44/76 strain (Day 335): number analyzed (Participants) | 127 | 64
  H44/76 strain (Day 335) | 99 [95.7 to 99.98] | 0 [0.0 to 5.6]
  5/99 strain (Day 1): number analyzed (Participants) | 141 | 72
  5/99 strain (Day 1) | 1 [0.02 to 3.9] | 0 [0.0 to 5.0]
  5/99 strain (Day 152): number analyzed (Participants) | 129 | 70
  5/99 strain (Day 152) | 100 [97.2 to 100] | 0 [0.0 to 5.1]
  5/99 strain (Day 305): number analyzed (Participants) | 135 | 70
  5/99 strain (Day 305) | 99 [94.8 to 99.82] | 1 [0.04 to 7.7]
  5/99 strain (Day 335): number analyzed (Participants) | 134 | 71
  5/99 strain (Day 335) | 99 [94.7 to 99.82] | 0 [0.0 to 5.1]
  M10713 strain (Day 1): number analyzed (Participants) | 121 | 64
  M10713 strain (Day 1) | 3 [0.9 to 8.2] | 8 [2.6 to 17.3]
  M10713 strain (Day 152): number analyzed (Participants) | 123 | 65
  M10713 strain (Day 152) | 49 [39.7 to 58.0] | 5 [1.0 to 12.9]
  M10713 strain (Day 305): number analyzed (Participants) | 130 | 65
  M10713 strain (Day 305) | 15 [9.7 to 22.8] | 3 [0.37 to 10.7]
  M10713 strain (Day 335): number analyzed (Participants) | 130 | 69
  M10713 strain (Day 335) | 77 [68.7 to 83.9] | 6 [1.6 to 14.2]
  NZ98/254 strain (Day 1) | 0 [0.0 to 2.5] | 0 [0.0 to 4.9]
  NZ98/254 strain (Day 152): number analyzed (Participants) | 135 | 71
  NZ98/254 strain (Day 152) | 59 [49.7 to 66.9] | 0 [0.0 to 5.1]
  NZ98/254 strain (Day 305): number analyzed (Participants) | 136 | 70
  NZ98/254 strain (Day 305) | 9 [4.6 to 14.9] | 0 [0.0 to 5.1]
  NZ98/254 strain (Day 335): number analyzed (Participants) | 136 | 71
  NZ98/254 strain (Day 335) | 86 [79.0 to 91.4] | 0 [0.0 to 5.1]

7. Secondary Outcome: Number of Subjects Reporting Solicited Local Adverse Events (AEs) After Receiving Bexsero® Vaccine With Routine Vaccine or Routine Vaccines Alone, at 2, 4, 6 and 12 Months of Age.
Description: Number of subjects reporting solicited local AEs following concomitant administration of Bexsero® vaccine with routine vaccines (Infanrix-IPV + Hib®, Prevenar-13® and Engerix-B® at 2, 4 and 6 months of age and Priorix® and Varilrix® at 12 months of age)compared to when only routine vaccines were administered alone at 2,4,6 and 12 months. Solicited local symptoms assessed were Erythema, Induration, Swelling and Tenderness.
Time Frame: From day 1 (6 hours) to day 7 after each vaccination (1st, 2nd, 3rd and 4th vaccination)
Population: Analysis was done on Safety set population (solicited AEs).The safety set population (solicited AEs) included all subjects in the Exposed Population who provided postvaccination reactogenicity data.
Measure: Number; unit: Number of participants
Arm/Group | Bexsero + Routine Group | Routine Group
Number analyzed (Participants) | 148 | 73
Number of participants
  Any Erythema (1st Bexsero®): number analyzed (Participants) | 148 | 0
  Any Erythema (1st Bexsero®) | 54 |
  Grade 3 Erythema (1st Bexsero®): number analyzed (Participants) | 148 | 0
  Grade 3 Erythema (1st Bexsero®) | 0 |
  Any Swelling (1st Bexsero®): number analyzed (Participants) | 146 | 0
  Any Swelling (1st Bexsero®) | 34 |
  Grade 3 Swelling (1st Bexsero®): number analyzed (Participants) | 146 | 0
  Grade 3 Swelling (1st Bexsero®) | 0 |
  Any Induration (1st Bexsero®): number analyzed (Participants) | 147 | 0
  Any Induration (1st Bexsero®) | 63 |
  Grade 3 Induration (1st Bexsero®): number analyzed (Participants) | 147 | 0
  Grade 3 Induration (1st Bexsero®) | 0 |
  Any Tenderness (1st Bexsero®): number analyzed (Participants) | 147 | 0
  Any Tenderness (1st Bexsero®) | 75 |
  Grade 3 Tenderness (1st Bexsero®): number analyzed (Participants) | 147 | 0
  Grade 3 Tenderness (1st Bexsero®) | 8 |
  Any Erythema (1st Infanrix-IPV + Hib®) | 26 | 3
  Grade 3 Erythema(1st Infanrix-IPV+Hib®) | 0 | 0
  Any Swelling (1st Infanrix-IPV + Hib®) | 15 | 3
  Grade 3 Swelling(1st Infanrix-IPV+Hib®) | 0 | 0
  Any Tenderness (1st Infanrix-IPV + Hib®): number analyzed (Participants) | 146 | 73
  Any Tenderness (1st Infanrix-IPV + Hib®) | 45 | 12
  Grade 3Tenderness(1st Infanrix-IPV+Hib®): number analyzed (Participants) | 146 | 73
  Grade 3Tenderness(1st Infanrix-IPV+Hib®) | 2 | 0
  Any Induration(1st Infanrix-IPV + Hib®) | 23 | 11
  Grade 3Induration(1st Infanrix-IPV+Hib®) | 0 | 0
  Any Erythema (1st Prevenar-13®) | 26 | 9
  Grade 3 Erythema (1st Prevenar-13®) | 0 | 0
  Any Induration (1st Prevenar-13®) | 29 | 15
  Grade 3 Induration (1st Prevenar-13®) | 0 | 0
  Any Swelling (1st Prevenar-13®) | 11 | 4
  Grade 3 Swelling (1st Prevenar-13®) | 0 | 0
  Any Tenderness (1st Prevenar-13®): number analyzed (Participants) | 147 | 73
  Any Tenderness (1st Prevenar-13®) | 50 | 12
  Grade 3 Tenderness (1st Prevenar-13®): number analyzed (Participants) | 147 | 73
  Grade 3 Tenderness (1st Prevenar-13®) | 3 | 0
  Any Erythema (2nd Bexsero®): number analyzed (Participants) | 140 | 0
  Any Erythema (2nd Bexsero®) | 59 |
  Grade 3 Erythema (2nd Bexsero®): number analyzed (Participants) | 140 | 0
  Grade 3 Erythema (2nd Bexsero®) | 0 |
  Any Swelling (2nd Bexsero®): number analyzed (Participants) | 140 | 0
  Any Swelling (2nd Bexsero®) | 35 |
  Grade 3 Swelling (2nd Bexsero®): number analyzed (Participants) | 140 | 0
  Grade 3 Swelling (2nd Bexsero®) | 0 |
  Any Induration (2nd Bexsero®): number analyzed (Participants) | 140 | 0
  Any Induration (2nd Bexsero®) | 51 |
  Grade 3 Induration (2nd Bexsero®): number analyzed (Participants) | 140 | 0
  Grade 3 Induration (2nd Bexsero®) | 0 |
  Any Tenderness (2nd Bexsero®): number analyzed (Participants) | 140 | 0
  Any Tenderness (2nd Bexsero®) | 67 |
  Grade 3 Tenderness (2nd Bexsero®): number analyzed (Participants) | 140 | 0
  Grade 3 Tenderness (2nd Bexsero®) | 5 |
  Any Erythema (2nd Infanrix-IPV + Hib®): number analyzed (Participants) | 140 | 72
  Any Erythema (2nd Infanrix-IPV + Hib®) | 39 | 12
  Grade 3 Erythema(2nd Infanrix-IPV+Hib®): number analyzed (Participants) | 140 | 72
  Grade 3 Erythema(2nd Infanrix-IPV+Hib®) | 0 | 0
  Any Swelling (2nd Infanrix-IPV + Hib®): number analyzed (Participants) | 140 | 72
  Any Swelling (2nd Infanrix-IPV + Hib®) | 18 | 6
  Grade 3 Swelling(2nd Infanrix-IPV+Hib®): number analyzed (Participants) | 140 | 72
  Grade 3 Swelling(2nd Infanrix-IPV+Hib®) | 0 | 0
  Any Induration (2nd Infanrix-IPV + Hib®): number analyzed (Participants) | 140 | 72
  Any Induration (2nd Infanrix-IPV + Hib®) | 23 | 16
  Grade 3Induration(2nd Infanrix-IPV+Hib®): number analyzed (Participants) | 140 | 72
  Grade 3Induration(2nd Infanrix-IPV+Hib®) | 0 | 0
  Any Tenderness (2nd Infanrix-IPV + Hib®): number analyzed (Participants) | 140 | 72
  Any Tenderness (2nd Infanrix-IPV + Hib®) | 45 | 10
  Grade 3Tenderness(2nd Infanrix-IPV+Hib®): number analyzed (Participants) | 140 | 72
  Grade 3Tenderness(2nd Infanrix-IPV+Hib®) | 3 | 0
  Any Erythema (2nd Prevenar-13®): number analyzed (Participants) | 140 | 72
  Any Erythema (2nd Prevenar-13®) | 35 | 12
  Grade 3 Erythema (2nd Prevenar-13®): number analyzed (Participants) | 140 | 72
  Grade 3 Erythema (2nd Prevenar-13®) | 0 | 0
  Any Induration (2nd Prevenar-13®): number analyzed (Participants) | 140 | 72
  Any Induration (2nd Prevenar-13®) | 18 | 8
  Grade 3 Induration (2nd Prevenar-13®): number analyzed (Participants) | 140 | 72
  Grade 3 Induration (2nd Prevenar-13®) | 0 | 0
  Any Swelling (2nd Prevenar-13®): number analyzed (Participants) | 140 | 72
  Any Swelling (2nd Prevenar-13®) | 12 | 6
  Grade 3 Swelling (2nd Prevenar-13®): number analyzed (Participants) | 140 | 72
  Grade 3 Swelling (2nd Prevenar-13®) | 0 | 0
  Any Tenderness (2nd Prevenar-13®): number analyzed (Participants) | 140 | 72
  Any Tenderness (2nd Prevenar-13®) | 44 | 9
  Grade 3 Tenderness (2nd Prevenar-13®): number analyzed (Participants) | 140 | 72
  Grade 3 Tenderness (2nd Prevenar-13®) | 3 | 0
  Any Erythema (3rd Engerix-B®): number analyzed (Participants) | 138 | 72
  Any Erythema (3rd Engerix-B®) | 33 | 12
  Grade 3 Erythema (3rd Engerix-B®): number analyzed (Participants) | 138 | 72
  Grade 3 Erythema (3rd Engerix-B®) | 0 | 0
  Any Induration (3rd Engerix-B®): number analyzed (Participants) | 137 | 72
  Any Induration (3rd Engerix-B®) | 33 | 17
  Grade 3 Induration (3rd Engerix-B®): number analyzed (Participants) | 137 | 72
  Grade 3 Induration (3rd Engerix-B®) | 0 | 0
  Any Swelling (3rd Engerix-B®): number analyzed (Participants) | 138 | 71
  Any Swelling (3rd Engerix-B®) | 25 | 6
  Grade 3 Swelling (3rd Engerix-B®): number analyzed (Participants) | 138 | 71
  Grade 3 Swelling (3rd Engerix-B®) | 0 | 0
  Any Tenderness (3rd Engerix-B®): number analyzed (Participants) | 138 | 72
  Any Tenderness (3rd Engerix-B®) | 45 | 7
  Grade 3 Tenderness (3rd Engerix-B®): number analyzed (Participants) | 138 | 72
  Grade 3 Tenderness (3rd Engerix-B®) | 3 | 0
  Any Erythema (3rd Bexsero®): number analyzed (Participants) | 138 | 0
  Any Erythema (3rd Bexsero®) | 55 |
  Grade 3 Erythema (3rd Bexsero®): number analyzed (Participants) | 138 | 0
  Grade 3 Erythema (3rd Bexsero®) | 0 |
  Any Induration (3rd Bexsero®): number analyzed (Participants) | 138 | 0
  Any Induration (3rd Bexsero®) | 57 |
  Grade 3 Induration (3rd Bexsero®): number analyzed (Participants) | 138 | 0
  Grade 3 Induration (3rd Bexsero®) | 0 |
  Any Swelling (3rd Bexsero®): number analyzed (Participants) | 138 | 0
  Any Swelling (3rd Bexsero®) | 49 |
  Grade 3 Swelling (3rd Bexsero®): number analyzed (Participants) | 138 | 0
  Grade 3 Swelling (3rd Bexsero®) | 0 |
  Any Tenderness (3rd Bexsero®): number analyzed (Participants) | 138 | 0
  Any Tenderness (3rd Bexsero®) | 68 |
  Grade 3 Tenderness (3rd Bexsero®): number analyzed (Participants) | 138 | 0
  Grade 3 Tenderness (3rd Bexsero®) | 6 |
  Any Swelling (3rd Infanrix-IPV+Hib®): number analyzed (Participants) | 148 | 72
  Any Swelling (3rd Infanrix-IPV+Hib®) | 20 | 10
  Grade 3 Swelling (3rd Infanrix-IPV+Hib®): number analyzed (Participants) | 138 | 72
  Grade 3 Swelling (3rd Infanrix-IPV+Hib®) | 0 | 0
  Any Erythema (3rd Infanrix-IPV+Hib®): number analyzed (Participants) | 137 | 72
  Any Erythema (3rd Infanrix-IPV+Hib®) | 28 | 15
  Grade 3 Erythema (3rd Infanrix-IPV+Hib®): number analyzed (Participants) | 137 | 72
  Grade 3 Erythema (3rd Infanrix-IPV+Hib®) | 0 | 0
  Any Induration(3rd Infanrix-IPV+Hib®): number analyzed (Participants) | 138 | 72
  Any Induration(3rd Infanrix-IPV+Hib®) | 25 | 16
  Grade 3Induration(3rd Infanrix-IPV+Hib®): number analyzed (Participants) | 138 | 72
  Grade 3Induration(3rd Infanrix-IPV+Hib®) | 0 | 0
  Any Tenderness (3rd Infanrix-IPV+ Hib®): number analyzed (Participants) | 138 | 72
  Any Tenderness (3rd Infanrix-IPV+ Hib®) | 42 | 8
  Grade 3Tenderness(3rd Infanrix-IPV+Hib®): number analyzed (Participants) | 138 | 72
  Grade 3Tenderness(3rd Infanrix-IPV+Hib®) | 2 | 0
  Any Erythema (3rd Prevenar-13®): number analyzed (Participants) | 138 | 72
  Any Erythema (3rd Prevenar-13®) | 27 | 12
  Grade 3 Erythema (3rd Prevenar-13®): number analyzed (Participants) | 138 | 72
  Grade 3 Erythema (3rd Prevenar-13®) | 0 | 0
  Any Induration (3rd Prevenar-13®): number analyzed (Participants) | 138 | 72
  Any Induration (3rd Prevenar-13®) | 21 | 11
  Grade 3 Induration (3rd Prevenar-13®): number analyzed (Participants) | 138 | 72
  Grade 3 Induration (3rd Prevenar-13®) | 0 | 0
  Any Swelling (3rd Prevenar-13®): number analyzed (Participants) | 138 | 72
  Any Swelling (3rd Prevenar-13®) | 17 | 4
  Grade 3 Swelling (3rd Prevenar-13®): number analyzed (Participants) | 138 | 72
  Grade 3 Swelling (3rd Prevenar-13®) | 0 | 0
  Any Tenderness (3rd Prevenar-13®): number analyzed (Participants) | 138 | 72
  Any Tenderness (3rd Prevenar-13®) | 45 | 9
  Grade 3 Tenderness (3rd Prevenar-13®): number analyzed (Participants) | 138 | 72
  Grade 3 Tenderness (3rd Prevenar-13®) | 3 | 0
  Any Erythema (4th Bexsero®): number analyzed (Participants) | 136 | 0
  Any Erythema (4th Bexsero®) | 53 |
  Grade 3 Erythema (4th Bexsero®): number analyzed (Participants) | 136 | 0
  Grade 3 Erythema (4th Bexsero®) | 0 |
  Any Swelling (4th Bexsero®): number analyzed (Participants) | 135 | 0
  Any Swelling (4th Bexsero®) | 44 |
  Grade 3 Swelling (4th Bexsero®): number analyzed (Participants) | 135 | 0
  Grade 3 Swelling (4th Bexsero®) | 0 |
  Any Induration (4th Bexsero®): number analyzed (Participants) | 136 | 0
  Any Induration (4th Bexsero®) | 56 |
  Grade 3 Induration(4th Bexsero®): number analyzed (Participants) | 136 | 0
  Grade 3 Induration(4th Bexsero®) | 0 |
  Any Tenderness (4th Bexsero®): number analyzed (Participants) | 136 | 0
  Any Tenderness (4th Bexsero®) | 66 |
  Grade 3 Tenderness (4th Bexsero®): number analyzed (Participants) | 136 | 0
  Grade 3 Tenderness (4th Bexsero®) | 6 |
  Any Erythema (4th Priorix®): number analyzed (Participants) | 137 | 72
  Any Erythema (4th Priorix®) | 24 | 13
  Grade 3 Erythema (4th Priorix®): number analyzed (Participants) | 137 | 72
  Grade 3 Erythema (4th Priorix®) | 0 | 0
  Any Induration (4th Priorix®): number analyzed (Participants) | 137 | 72
  Any Induration (4th Priorix®) | 15 | 6
  Grade 3 Induration (4th Priorix®): number analyzed (Participants) | 137 | 72
  Grade 3 Induration (4th Priorix®) | 0 | 0
  Any Swelling (4th Priorix®): number analyzed (Participants) | 137 | 72
  Any Swelling (4th Priorix®) | 19 | 4
  Grade 3 Swelling (4th Priorix®): number analyzed (Participants) | 137 | 72
  Grade 3 Swelling (4th Priorix®) | 0 | 0
  Any Tenderness (4th Priorix®): number analyzed (Participants) | 137 | 72
  Any Tenderness (4th Priorix®) | 37 | 6
  Grade 3 Tenderness (4th Priorix®): number analyzed (Participants) | 137 | 72
  Grade 3 Tenderness (4th Priorix®) | 3 | 0
  Any Erythema (4th Varilrix®): number analyzed (Participants) | 137 | 72
  Any Erythema (4th Varilrix®) | 32 | 14
  Grade 3 Erythema (4th Varilrix®): number analyzed (Participants) | 137 | 72
  Grade 3 Erythema (4th Varilrix®) | 0 | 0
  Any Induration (4th Varilrix®): number analyzed (Participants) | 137 | 72
  Any Induration (4th Varilrix®) | 14 | 7
  Grade 3 Induration (4th Varilrix®): number analyzed (Participants) | 137 | 72
  Grade 3 Induration (4th Varilrix®) | 0 | 0
  Any Swelling (4th Varilrix®): number analyzed (Participants) | 137 | 72
  Any Swelling (4th Varilrix®) | 21 | 6
  Grade 3 Swelling (4th Varilrix®): number analyzed (Participants) | 137 | 72
  Grade 3 Swelling (4th Varilrix®) | 0 | 0
  Any Tenderness (4th Varilrix®): number analyzed (Participants) | 137 | 72
  Any Tenderness (4th Varilrix®) | 41 | 5
  Grade 3 Tenderness (4th Varilrix®): number analyzed (Participants) | 137 | 72
  Grade 3 Tenderness (4th Varilrix®) | 3 | 0

8. Secondary Outcome: Number of Subjects Reporting Solicited Systemic Adverse Events (AEs) After Receiving Bexsero® Vaccine With Routine Vaccine or Routine Vaccines Alone, at 2, 4, 6 and 12 Months of Age.
Description: Number of subjects reporting solicited systemic AEs following concomitant administration of Bexsero® vaccine with routine vaccines (Infanrix-IPV + Hib®, Prevenar-13® and Engerix-B® at 2, 4 and 6 months of age and Priorix® and Varilrix® at 12 months of age) compared to when only routine vaccines were alone, at 2, 4, 6 and 12 months. Systemic solicited symptoms assessed were Change in Eating Habits, Diarrhea, Irritability, Persistent Crying, Rash, Sleepiness, Vomiting and Fever (body temperature ≥ 38.0 °C)
Time Frame: From day 1 (6 hours) to day 7 after each vaccination
Population: as for outcome 7
Measure: Number; unit: Number of participants
Arm/Group | Bexsero + Routine Group | Routine Group
Number analyzed (Participants) | 148 | 73
Number of participants
  Any Change in Eating Habits (1st vacc) | 92 | 26
  Grade3 Change in Eating Habits(1st vacc) | 0 | 0
  Any Change in Eating Habits (2nd vacc): number analyzed (Participants) | 140 | 72
  Any Change in Eating Habits (2nd vacc) | 72 | 21
  Grade3 Change in Eating Habits(2nd vacc): number analyzed (Participants) | 140 | 72
  Grade3 Change in Eating Habits(2nd vacc) | 2 | 0
  Any Change in Eating Habits (3rd vacc): number analyzed (Participants) | 138 | 72
  Any Change in Eating Habits (3rd vacc) | 72 | 17
  Grade3 Change in Eating Habits(3rd vacc): number analyzed (Participants) | 138 | 72
  Grade3 Change in Eating Habits(3rd vacc) | 1 | 0
  Any Diarrhea (1st vacc) | 28 | 8
  Grade 3 Diarrhea (1st vacc) | 2 | 1
  Any Diarrhea (2nd vacc): number analyzed (Participants) | 140 | 72
  Any Diarrhea (2nd vacc) | 30 | 9
  Grade 3 Diarrhea (2nd vacc): number analyzed (Participants) | 140 | 72
  Grade 3 Diarrhea (2nd vacc) | 1 | 0
  Any Diarrhea (3rd vacc): number analyzed (Participants) | 138 | 72
  Any Diarrhea (3rd vacc) | 19 | 4
  Grade 3 Diarrhea (3rd vacc): number analyzed (Participants) | 138 | 72
  Grade 3 Diarrhea (3rd vacc) | 0 | 0
  Any Irritability (1st vacc) | 111 | 32
  Grade 3 Irritability (1st vacc) | 3 | 0
  Any Irritability (2nd vacc): number analyzed (Participants) | 140 | 72
  Any Irritability (2nd vacc) | 90 | 31
  Grade 3 Irritability (2nd vacc): number analyzed (Participants) | 140 | 72
  Grade 3 Irritability (2nd vacc) | 5 | 0
  Any Irritability (3rd vacc): number analyzed (Participants) | 138 | 72
  Any Irritability (3rd vacc) | 94 | 28
  Grade 3 Irritability (3rd vacc): number analyzed (Participants) | 138 | 72
  Grade 3 Irritability (3rd vacc) | 3 | 1
  Any Persistent Crying (1st vacc) | 96 | 30
  Grade 3 Persistent Crying (1st vacc) | 5 | 0
  Any Persistent Crying (2nd vacc): number analyzed (Participants) | 140 | 72
  Any Persistent Crying (2nd vacc) | 82 | 23
  Grade 3 Persistent Crying (2nd vacc): number analyzed (Participants) | 140 | 72
  Grade 3 Persistent Crying (2nd vacc) | 5 | 0
  Any Persistent Crying (3rd vacc): number analyzed (Participants) | 138 | 72
  Any Persistent Crying (3rd vacc) | 72 | 28
  Grade 3 Persistent Crying (3rd vacc): number analyzed (Participants) | 138 | 72
  Grade 3 Persistent Crying (3rd vacc) | 3 | 0
  Any Rash (1st vacc) | 18 | 4
  Grade 3 Rash (1st vacc) | 0 | 0
  Any Rash (2nd vacc): number analyzed (Participants) | 140 | 72
  Any Rash (2nd vacc) | 18 | 8
  Grade 3 Rash (2nd vacc): number analyzed (Participants) | 140 | 72
  Grade 3 Rash (2nd vacc) | 0 | 1
  Any Rash (3rd vacc): number analyzed (Participants) | 138 | 72
  Any Rash (3rd vacc) | 16 | 4
  Grade 3 Rash (3rd vacc): number analyzed (Participants) | 138 | 72
  Grade 3 Rash (3rd vacc) | 1 | 0
  Any Sleepiness (1st vacc) | 79 | 33
  Grade 3 Sleepiness (1st vacc) | 0 | 1
  Any Sleepiness (2nd vacc): number analyzed (Participants) | 140 | 72
  Any Sleepiness (2nd vacc) | 66 | 21
  Grade 3 Sleepiness (2nd vacc): number analyzed (Participants) | 140 | 72
  Grade 3 Sleepiness (2nd vacc) | 0 | 0
  Any Sleepiness (3rd vacc): number analyzed (Participants) | 138 | 72
  Any Sleepiness (3rd vacc) | 49 | 13
  Grade 3 Sleepiness (3rd vacc): number analyzed (Participants) | 138 | 72
  Grade 3 Sleepiness (3rd vacc) | 0 | 0
  Any Vomiting (1st vacc) | 21 | 6
  Grade 3 Vomiting (1st vacc) | 0 | 0
  Any Vomiting (2nd vacc): number analyzed (Participants) | 140 | 72
  Any Vomiting (2nd vacc) | 16 | 9
  Grade 3 Vomiting (2nd vacc): number analyzed (Participants) | 140 | 72
  Grade 3 Vomiting (2nd vacc) | 0 | 0
  Any Vomiting (3rd vacc): number analyzed (Participants) | 138 | 72
  Any Vomiting (3rd vacc) | 15 | 7
  Grade 3 Vomiting (3rd vacc): number analyzed (Participants) | 138 | 72
  Grade 3 Vomiting (3rd vacc) | 0 | 0
  Fever (1st vacc) | 71 | 11
  Fever (2nd vacc): number analyzed (Participants) | 140 | 71
  Fever (2nd vacc) | 72 | 11
  Fever (3rd vacc): number analyzed (Participants) | 138 | 72
  Fever (3rd vacc) | 68 | 12
  Any Change in Eating Habits (4th vacc): number analyzed (Participants) | 137 | 72
  Any Change in Eating Habits (4th vacc) | 58 | 19
  Grade3 Change in Eating Habits(4th vacc): number analyzed (Participants) | 137 | 72
  Grade3 Change in Eating Habits(4th vacc) | 2 | 1
  Any Diarrhea (4th vacc): number analyzed (Participants) | 137 | 72
  Any Diarrhea (4th vacc) | 27 | 10
  Grade 3 Diarrhea (4th vacc): number analyzed (Participants) | 137 | 72
  Grade 3 Diarrhea (4th vacc) | 1 | 0
  Any Irritability (4th vacc): number analyzed (Participants) | 137 | 72
  Any Irritability (4th vacc) | 71 | 16
  Grade 3 Irritability (4th vacc): number analyzed (Participants) | 137 | 72
  Grade 3 Irritability (4th vacc) | 2 | 0
  Any Persistent Crying (4th vacc): number analyzed (Participants) | 137 | 72
  Any Persistent Crying (4th vacc) | 58 | 15
  Grade 3 Persistent Crying (4th vacc): number analyzed (Participants) | 137 | 72
  Grade 3 Persistent Crying (4th vacc) | 0 | 1
  Any Rash (4th vacc): number analyzed (Participants) | 137 | 72
  Any Rash (4th vacc) | 25 | 9
  Grade 3 Rash (4th vacc): number analyzed (Participants) | 137 | 72
  Grade 3 Rash (4th vacc) | 1 | 0
  Any Sleepiness (4th vacc): number analyzed (Participants) | 137 | 72
  Any Sleepiness (4th vacc) | 36 | 9
  Grade 3 Sleepiness (4th vacc): number analyzed (Participants) | 137 | 72
  Grade 3 Sleepiness (4th vacc) | 0 | 0
  Any Vomiting (4th vacc): number analyzed (Participants) | 137 | 72
  Any Vomiting (4th vacc) | 10 | 6
  Grade 3 Vomiting (4th vacc): number analyzed (Participants) | 137 | 72
  Grade 3 Vomiting (4th vacc) | 0 | 0
  Fever (4th vacc): number analyzed (Participants) | 137 | 72
  Fever (4th vacc) | 60 | 6
  Lymphadenopathy (4th vacc): number analyzed (Participants) | 137 | 72
  Lymphadenopathy (4th vacc) | 1 | 1

9. Secondary Outcome: Number of Subjects Reporting Solicited Systemic AEs After Receiving Priorix® and Varilrix® Routine Vaccines (With and Without Bexsero® Vaccine) at 12 Months of Age.
Description: Number of subjects who reported solicited systemic AEs reported after the administration of Varilrix® and Priorix® vaccines (with and without Bexsero® vaccine) at 12 months of age. Solicited systemic AEs assessed were Rash, Lymphadenopathy and Fever. This analysis was conducted for a prolonged period of 28 Days following Varilrix® and Priorix® administration.
Time Frame: From Day 1 to Day 28 after vaccination
Population: as for outcome 7
Measure: Number; unit: Number of participants
Arm/Group | Bexsero + Routine Group | Routine Group
Number analyzed (Participants) | 137 | 72
Number of participants
  Any Rash (4th vacc) | 50 | 24
  Grade 3 rash (4th vacc) | 5 | 5
  Lymphadenopathy (4th vacc) | 34 | 21
  Fever (temperature ≥ 38.0°C) | 91 | 33
  Grade 3 fever (temperature ≥ 40.0°C) | 2 | 5

10. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events After Receiving Bexsero® Vaccination With Routine Vaccines
Description: Number of subjects reporting any unsolicited AEs following concomitant administration of Bexsero® vaccine with routine vaccines (Infanrix-IPV + Hib®, Prevenar-13®, Engerix-B® or Priorix® and Varilrix®) compared to when only routine vaccines were administered alone.
Time Frame: From day 1 to day 7 after each vaccination
Population: Analysis was done on Safety set population (unsolicited AEs). The safety set population (unsolicited AEs) included all subjects in the Exposed Population who had postvaccination unsolicited AE records.
Measure: Number; unit: Number of subjects
Arm/Group | Bexsero + Routine Group | Routine Group
Number analyzed (Participants) | 145 | 72
Number of subjects
  Any AEs (1st vacc) | 46 | 8
  At least possible related AEs (1st vacc) | 35 | 6
  Any AEs (2nd vacc): number analyzed (Participants) | 141 | 72
  Any AEs (2nd vacc) | 30 | 7
  At least possible related AEs (2nd vacc): number analyzed (Participants) | 141 | 72
  At least possible related AEs (2nd vacc) | 22 | 5
  Any AEs (3rd vacc): number analyzed (Participants) | 138 | 72
  Any AEs (3rd vacc) | 51 | 18
  At least possible related AEs (3rd vacc): number analyzed (Participants) | 138 | 72
  At least possible related AEs (3rd vacc) | 45 | 7
  Any AEs (booster): number analyzed (Participants) | 137 | 72
  Any AEs (booster) | 43 | 9
  At least possible related AEs (booster): number analyzed (Participants) | 137 | 72
  At least possible related AEs (booster) | 37 | 4

11. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs), Medically Attended AEs (MAEs) and AEs Leading to Premature Withdrawal and Death and AEs Leading to Hospitalization.
Description: Number of subjects reporting SAEs, medically attended AEs and AEs leading to premature withdrawal from the study and leading to death and AEs leading to hospitalization following concomitant administration of Bexsero® vaccine with routine vaccines (Infanrix-IPV + Hib®, Prevenar-13®, Engerix-B®, Priorix® and Varilrix®) compared to when only routine vaccines were administered alone. SAEs assessed included medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Possibly or probably related SAE were SAEs assessed by the investigator as related to the vaccination. Medically attended AEs were events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason.
Time Frame: Throughout the study period (Day 1 to Day 335)
Population: as for outcome 10
Measure: Number; unit: Number of participants
Arm/Group | Bexsero + Routine Group | Routine Group
Number analyzed (Participants) | 145 | 72
Number of participants
  Any SAEs | 13 | 8
  At least possible related SAEs | 0 | 0
  AEs resulting in premature withdrawal | 4 | 0
  AEs leading to hospitalization | 13 | 8
  Medically attended AEs | 131 | 66
  AEs leading to death | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local AEs and systemic symptoms: from Day 1 to Day 7 after each vaccination; Unsolicited AEs and SAEs: throughout the study period (from Day 1 to Day 335).
Description: Serious adverse events were analysed based on the unsolicited safety set and other adverse events were analysed based on the overall safety set. Therefore, the number of participants at risk in the serious adverse events are lesser compared to the number of participants at risk in the other adverse events.
Arm/Group | Bexsero + Routine Group | Routine Group
All-Cause Mortality (participants affected / at risk) | 0/148 | 0/73
Serious Adverse Events (participants affected / at risk) | 13/145 | 8/72
Other Adverse Events (participants affected / at risk) | 148/148 | 72/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bexsero + Routine Group (N=145) | Routine Group (N=72)
Kawasaki's disease (Vascular disorders) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Bronchiolitis (Infections and infestations) | 3 | 1
Urinary tract infection (Infections and infestations) | 4 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 2 | 0
Otitis media acute (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0
Croup infectious (Infections and infestations) | 0 | 1
Exanthema subitum (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Pyuria (Infections and infestations) | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 1
Salmonella bacteraemia (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bexsero + Routine Group (N=148) | Routine Group (N=73)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Somnolence (Nervous system disorders) | 111 | 45
Pyrexia (General disorders) | 134 | 51
Crying (General disorders) | 124 | 50
Injection site erythema (General disorders) | 113 | 35
Injection site pain (General disorders) | 121 | 27
Injection site induration (General disorders) | 105 | 39
Injection site swelling (General disorders) | 89 | 24
Irritability (Psychiatric disorders) | 127 | 50
Eating disorder (Psychiatric disorders) | 125 | 43
Diarrhoea (Gastrointestinal disorders) | 72 | 29
Vomiting (Gastrointestinal disorders) | 45 | 16
Rash (Skin and subcutaneous tissue disorders) | 72 | 30
Eczema (Skin and subcutaneous tissue disorders) | 17 | 5
Dermatitis (Skin and subcutaneous tissue disorders) | 15 | 4
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 8 | 5
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 7 | 6
Nasopharyngitis (Infections and infestations) | 86 | 45
Upper respiratory tract infection (Infections and infestations) | 42 | 16
Bronchiolitis (Infections and infestations) | 9 | 4
Exanthema subitum (Infections and infestations) | 9 | 6
Conjunctivitis (Infections and infestations) | 5 | 4
Pharyngitis (Infections and infestations) | 5 | 4
Tonsillitis (Infections and infestations) | 4 | 4
Gastroenteritis (Infections and infestations) | 14 | 12
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 34 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.